CLINICAL TRIAL: NCT07181330
Title: Retrospective Clinical Validation of the SE-SPTM-PCR Platform for Hcmv-miR-UL22A-5p Detection in Monitoring Cytomegalovirus Infection After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Clinical Performance of SE-SPTM-PCR in Detecting Hcmv-miR-UL22A-5p After Hematopoietic Stem Cell Transplantation
Acronym: SESPTM-CMV
Status: Completed | Type: Observational
Sponsor: Ting YANG (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Prof., Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: FMU-XMU-SESPTM-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections; Hematopoietic Stem Cell Transplantation (HSCT); CMV Reactivation; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION
Keywords: Cytomegalovirus; hcmv-miR-UL22A-5p; CMV reactivation; microRNA biomarker; miRNA detection; SE-SPTM-PCR; Hematopoietic Stem Cell Transplantation; Allogeneic HSCT; Liquid biopsy; Retrospective study; qPCR; Viral monitoring; Transplant infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived human plasma samples will be retained for analysis. The samples were collected from patients who underwent allogeneic hematopoietic stem cell transplantation. Each sample contains circulating RNA, including viral microRNAs such as hcmv-miR-UL22A-5p. All specimens are de-identified and stored in a coded format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSCT Patient Group: This group includes patients who underwent allogeneic hematopoietic stem cell transplantation (HSCT). Archived plasma samples from these patients are used to evaluate the performance of the SE-SPTM-PCR platform for detecting hcmv-miR-UL22A-5p. Each sample has a corresponding CMV DNA test result, which serves as the reference standard for assessing the diagnostic accuracy of the microRNA-based detection method.
  Interventions: Diagnostic Test: SE-SPTM-PCR microRNA assay

INTERVENTIONS:
Diagnostic Test: SE-SPTM-PCR microRNA assay — SE-SPTM-PCR (Selective Enrichment and Specific Probe Terminal Mediated PCR) is a microRNA-based diagnostic assay designed to detect hcmv-miR-UL22A-5p in human plasma. In this retrospective observational study, the assay is used on archived plasma samples collected from patients who underwent allogeneic hematopoietic stem cell transplantation (HSCT). The purpose is to evaluate the diagnostic performance of this method in identifying CMV reactivation, compared to standard CMV DNA qPCR testing. This test was not assigned or administered as part of patient care but is the primary focus of retrospective laboratory analysis.
  Other Names: SE-SPTM-PCR; Selective Enrichment and Specific Probe Terminal Mediated PCR; hcmv-miR-UL22A-5p assay; microRNA-based CMV test; HSCT CMV miRNA detection

SUMMARY:
This study aims to evaluate the clinical performance of a novel microRNA-based detection platform, SE-SPTM-PCR, for identifying cytomegalovirus (CMV) infection after allogeneic hematopoietic stem cell transplantation (HSCT). Specifically, the study retrospectively analyzes plasma samples to determine whether hcmv-miR-UL22A-5p can serve as a sensitive and specific biomarker for CMV reactivation. Results will be compared to traditional CMV DNA testing methods.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) reactivation is a frequent and serious complication after allogeneic hematopoietic stem cell transplantation (HSCT), potentially leading to CMV disease, graft-versus-host disease, and increased transplant-related mortality. Early and accurate monitoring of CMV infection is critical for timely treatment.

Traditional CMV monitoring relies on the detection of CMV DNA in blood using quantitative PCR. However, this method may have limited sensitivity in early infection stages or low viral load situations. MicroRNAs encoded by CMV, such as hcmv-miR-UL22A-5p, are small non-coding RNAs released into circulation during viral activity and may serve as alternative biomarkers.

This study retrospectively evaluates a novel microRNA-based detection platform, SE-SPTM-PCR (Selective Enrichment and Specific Probe Terminal Mediated PCR), for its ability to detect hcmv-miR-UL22A-5p in plasma samples from HSCT recipients. The goal is to determine whether this method improves the sensitivity and specificity of CMV reactivation monitoring compared to standard CMV DNA testing.

Archived plasma samples from post-HSCT patients with known CMV DNA status (positive or negative) will be tested. The diagnostic performance of SE-SPTM-PCR will be assessed through ROC curve analysis, correlation with DNA viral load, and comparison of sensitivity and specificity.

Findings from this study may support the use of hcmv-miR-UL22A-5p as a more sensitive and stable biomarker for CMV reactivation, and promote the clinical application of SE-SPTM-PCR in transplant monitoring strategies.

ELIGIBILITY:
Inclusion Criteria:

Patients who received allogeneic hematopoietic stem cell transplantation (HSCT)

Availability of archived plasma samples collected within 100 days post-transplant

Documented CMV DNA testing results corresponding to the plasma sample

Age ≥ 18 years

Exclusion Criteria:

Lack of corresponding CMV DNA testing results

Inadequate volume or quality of archived plasma sample for analysis

Concurrent active infections with other viruses (e.g., EBV, HBV, HCV) at time of plasma collection

Patients who received investigational antiviral therapy within 2 weeks prior to sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent allogeneic hematopoietic stem cell transplantation (HSCT) and had archived plasma samples collected within 100 days after transplantation. All participants had corresponding cytomegalovirus (CMV) DNA testing results available. Samples were retrospectively analyzed to assess the diagnostic performance of hcmv-miR-UL22A-5p using the SE-SPTM-PCR platform.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of SE-SPTM-PCR for detecting CMV reactivation | through study completion, an average of 1 month
  The primary outcome is the area under the receiver operating characteristic (ROC) curve (AUC) of SE-SPTM-PCR detection of hcmv-miR-UL22A-5p in plasma, compared to CMV DNA qPCR as the reference standard. Sensitivity and specificity will also be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No